CLINICAL TRIAL: NCT00840541
Title: Observational Study of Type-2 Diabetic Subjects to Validate Diabetic Retinopathy Phenotypes
Brief Title: Phenotyping Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: CNTM018A
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DR: Type-2 diabetic subjects diagnosed with diabetic retinopathy (DR).

SUMMARY:
The purpose of this study is to validate and characterize phenotypes of diabetic retinopathy (DR) progression based on available clinical data (demographic, systemic and ophthalmic data).

DETAILED DESCRIPTION:
This study aims to validate and characterize phenotypes of diabetic retinopathy (DR) progression using ophthalmic and systemic data from type-2 diabetic subjects followed at the AIBILI Clinical Trial Center in the last 10 years.

Macular Edema (ME) development during the study period, mainly Clinically Significant ME (CSME) needing treatment, will be the primary indicator for DR progression. CSME will be considered as the primary end-point and will be used to identify phenotypes (and risk markers) of DR progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DR.
* Females or Males;
* Age over 18 years;
* Signed Informed Consent;
* Previous follow-up with regular systemic and ophthalmic assessments.

Exclusion Criteria:

* Cataract or other eye disease that may interfere with fundus examinations;
* Vitreous syneresis or posterior vitreous detachment;
* Dilatation of the pupil < 5 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type-2 diabetic subjects diagnosed with DR, followed regularly by their ophthalmologist at the AIBILI Clinical Trial Center, with a previous follow-up in which systemic data and ophthalmological examinations were performed regularly.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
CSME | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI - Clinical Trial Center, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Background] Cunha-Vaz J. Characterization and relevance of different diabetic retinopathy phenotypes. Dev Ophthalmol. 2007;39:13-30. doi: 10.1159/000098497. PMID 17245076
- See also: Related Info — http://www.aibili.pt